CLINICAL TRIAL: NCT00883571
Title: Comparative Study of the House Advancement Flap, Rhomboid Flap, and Y-V Anoplasty in Treatment of Anal Stenosis: A Prospective Randomized Study
Brief Title: Comparative Study of the House Advancement Flap, Rhomboid Flap, and Y-V Anoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Mohmed Youssef, MANSOURA UNIVERSITY
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: anal stenosis
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2009-12-29 (Estimated); Status verified 2009-04

CONDITIONS: Anal Stenosis
Keywords: anal stenosis; flaps; anoplasty
MeSH Terms: conditions — Anus, Imperforate | interventions — gene 11 protein, Rotavirus B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- house advancement flap (Active Comparator): house advancement flap
  Interventions: Procedure: house advancement flap group
- Rhomboid flap (Active Comparator): rhomboid flapa was incised in the ischiorectal fossa. Without undermining of its fatty base, the flap was then mobilized into the anal canal so that the tip could be sutured to the top of the strictured area using Vicryl 3/0 sutures
  Interventions: Procedure: Rhomboid flap GROUP
- Y-V anoplasty (Active Comparator): Y-V anoplasty
  Interventions: Procedure: Y-V anoplasty GROUP

INTERVENTIONS:
Procedure: house advancement flap group — A house flap of healthy tissue was incised to the depth of ischiorectal fat. The flap consisted of skin and subcutaneous tissue. The flap was sufficiently mobilized without undermining its fatty base containing perforating blood vessels. The flap should be loose and easily advanced into the anal canal. When the ''base'' of this house-shaped flap was advanced into the anal canal defect, it was fixed to the top of the excised area with 3/0 Vicryl sutures.
  Other Names: group 1
  Arms: house advancement flap
Procedure: Rhomboid flap GROUP — A rhomboid flap was incised in ischeorectal fossa and was mobilized without undermining of its fatty base into the anal canal so that the tip of rhomboid flap is sutured to the top of stricured area using vicryl 3/0.
  Other Names: Group 11
  Arms: Rhomboid flap
Procedure: Y-V anoplasty GROUP — Y-V anoplastyis performed by making a v shaped incision in the perianal skin posteriorly starting from the lower end of the wound resultant from excision of scared area. A V-shaped flap is then dissected with preservation fatty base .The V flap is then advanced into the anal canal so that its tip is sutured to the top of structured area using vicryel 3/0.
  Other Names: group 111
  Arms: Y-V anoplasty

SUMMARY:
This prospective randomized study included 60 consecutive patients suffering from anal stenosis in the period from April 2002 to December 2008. They admitted to colorectal surgery unit, Mansoura university hospital, Egypt. According to the classification proposed by Milson and Mazier(5), all patients had moderate to severe anal stenosis. There were 43 males and 17 female with a mean age 34 + 5.2 years ranging from 18 up to 63 years.

DETAILED DESCRIPTION:
Informed consent was obtained from all patients to be included in the study, after explanations the nature of the disease and possible treatment. This study was approved by local ethical committee.

The patients were then randomized into three groups. The randomization was achieved through computer-generated schedule and its results were sealed into 60 envelopes. The responsible surgeon opened randomly an envelop and, accordingly to the protocol.

Group 1: consists of 20 (14 males and 6 females) patients underwent house door flap.

Group II: consists of 20 patients (16 males and 4 females) underwent romboid flap.

Group III: consists of 20 patients underwent V-Y anoplasty (13 males and 7 females).

In group I: a house flap of healthy tissue was incised to the depth of ischiorectal fat. The flap consisted of skin and subcutaneous tissue. The flap was sufficiently mobilized without undermining its fatty base containing perforating blood vessels. The flap should be loose and easily advanced into the anal canal. When the ''base'' of this house-shaped flap was advanced into the anal canal defect, it was fixed to the top of the excised area with 3/0 Vicryl sutures.

In group II: a rhomboid flap was incised in ischiorectal fossa and was mobilized without undermining of its fatty base into the anal canal so that the tip of rhomboid flap is sutured to the top of strictured area using vicryl 3/0.

In group III: V-Y anoplasty is performed by making a v shaped incision in the perianal skin posteriorly starting from the lower end of the wound resultant from excision of scared area. A V-shaped flap is then dissected with preservation fatty base .The V flap is then advanced into the anal canal so that its tip is sutured to the top of structured area using vicryel 3/0.

Patients were discharged 48 hours after the procedure. A high-fiber diet combined with bulk laxatives with oral antibiotic coverage was recommended after discharge. After each bowel movement, cleansing of the operative site with a sitz bath or shower was prescribed.

Patients were discharged 48 hours after the procedure. A high-fiber diet combined with bulk laxatives with oral antibiotic coverage was recommended after discharge. After each bowel movement, cleansing of the operative site with a sitz bath or shower was prescribed.

The parameters investigated were time of relief of painful defecation, the straining severity, sensation of incomplete evacuation and need for laxative or enema. postoperative anal caliber, healing rate, recurrence, quality of life (QOL) was assessed with Gastrointestinal quality of life index (GIQLI) which is a relatively new and validated tool for measuring the QOL in patients with gastrointestinal diseases. The GIQLI developed by Eypasch and coworkers (6). The questionnaire comprises 36 multidimensional items covering symptoms and physical, emotional, and social dysfunction related to gastrointestinal diseases or their treatments. Each item is scored from 0 to 4 points. The GIQLI score is calculated by simple addition of all item scores so that an overall score of 0 would constitute the worst, while a score of 144 (36 X 4) represents the best possible result. It is also possible to evaluate the disease-specific, social, psychologic, and physical items as separate subgroups. The patients were asked to complete the GIQLI questionnaire at admission to the hospital and one year after surgery under the supervision of the same independent authors.

ELIGIBILITY:
Inclusion Criteria:

* ALL PATIENTS with anal stenosis

Exclusion Criteria:

* Pregnant female
* Malignant stenosis
* Associated anal pathology
* Anal stenosis with a anal diameter more than 20 mm

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2002-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
postoperative anal caliber | 1 year

SECONDARY OUTCOMES:
clinical improvement, complications, recurrence, patient satisfaction, postoperative incontinence, and quality of life | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: mohamed yousef, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Egypt

REFERENCES:
- [Result] Habr-Gama A, Sobrado CW, de Araujo SE, Nahas SC, Birbojm I, Nahas CS, Kiss DR. Surgical treatment of anal stenosis: assessment of 77 anoplasties. Clinics (Sao Paulo). 2005 Feb;60(1):17-20. doi: 10.1590/s1807-59322005000100005. Epub 2005 Mar 1. PMID 15838576
- [Result] Alver O, Ersoy YE, Aydemir I, Erguney S, Teksoz S, Apaydin B, Ertem M. Use of "house" advancement flap in anorectal diseases. World J Surg. 2008 Oct;32(10):2281-6. doi: 10.1007/s00268-008-9699-1. PMID 18679744
- [Result] Eypasch E, Williams JI, Wood-Dauphinee S, Ure BM, Schmulling C, Neugebauer E, Troidl H. Gastrointestinal Quality of Life Index: development, validation and application of a new instrument. Br J Surg. 1995 Feb;82(2):216-22. doi: 10.1002/bjs.1800820229. PMID 7749697
- See also: mansoura university hospital — http://www.mans.edu.eg/